CLINICAL TRIAL: NCT06171529
Title: Efficacy of a Single Injection of Connective Tissue Matrix for Post-Operative CMC Arthritis
Brief Title: Efficacy of a Single Injection of CTM for Post-Operative CMC Arthritis
Acronym: CTM CMC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Indiana Hand to Shoulder Center (Other)
Collaborators: CTM Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: IHTSC CTM Series HC22-3
Record Dates: First submitted 2023-12-01; First posted 2023-12-14 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2023-12

CONDITIONS: Osteoarthritis; Osteoarthritis Thumb Base Joint; Carpometacarpal Osteoarthritis; Thumb
MeSH Terms: conditions — Osteoarthritis | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: For patients who randomize to CTM: An unblinded IHTSC Fellow, nurse/PA, or OR staff will use a 3 or 5 cc syringe to draw up the CTM Flow material. A 23, or 20 gauge needle will be used to inject the CTM after arthroplasty and prior to closure of the capsule. To draw up the injection: allow the particulate to settle to the bottom and withdrawal fluid into the 3 or 5 cc syringe. It is ok if some particulate is drawn up into the syringe. 2cc of CTM will be injected into each patient.
  For patients who randomize to Saline: An unblinded IHTSC Fellow, nurse/PA, or OR staff will use a 3 or 5 cc syringe to draw up the saline. A 23 gauge needle will be used to inject the saline after arthroplasty and prior to closure of the capsule. 2cc of saline will be injected into each patient.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Placebo - Saline (Placebo Comparator): For patients who randomize to Saline: An unblinded IHTSC Fellow, nurse/PA, or OR staff will use a 3 or 5 cc syringe to draw up the saline. A 23 gauge needle will be used to inject the saline after arthroplasty and prior to closure of the capsule. 2cc of saline will be injected into each patient.
  Interventions: Other: Placebo
- Treatment - CTM (Experimental): For patients who randomize to CTM: An unblinded IHTSC Fellow, nurse/PA, or OR staff will use a 3 or 5 cc syringe to draw up the CTM Flow material. A 23, or 20 gauge needle will be used to inject the CTM after arthroplasty and prior to closure of the capsule. To draw up the injection: allow the particulate to settle to the bottom and withdrawal fluid into the 3 or 5 cc syringe. It is ok if some particulate is drawn up into the syringe. 2cc of CTM will be injected into each patient.
  Interventions: Device: CTM

INTERVENTIONS:
Device: CTM — CTM Flow is stored in 1cc vials and is stable at room temperature and does not need to be refrigerated. CTM Flow will be supplied to and stored at the IHTSC Beltway Surgery Center. Product will be stored at room temperature without continued temperature control. All product will be kept in the Beltway Surgery Center and will not be separated from the marketed non-study CTM. Treating Surgeons will remain blinded to the treatment group, but will ensure that only the injection is billed to patients and the CTM or saline are provided at no cost. Lexie Reissaus, CCRP will track drug accountability.
  Arms: Treatment - CTM
Other: Placebo — placebo/Saline control injection
  Other Names: Saline
  Arms: Placebo - Saline

SUMMARY:
The goal of this study is to determine the success rate of a single Carpometacarpal (CMC) thumb injection after arthroplasty surgery for primary osteoarthritis of the CMC joint.

DETAILED DESCRIPTION:
CTM Biomedical markets and distributes decellularized particulate human placental connective-tissue matrix products, intended solely for homologous use to supplement or replace damaged or inadequate connective-tissue. These are structural tissue allografts processed according to the criteria contained in 21CFR 1271.10(a) for regulation solely under section 361 of the Public Health Service Act. CTM Flow is decellularized particulate human placental connective-tissue matrix provided in a vial.

Postoperative pain after basilar thumb arthritis reconstruction is often quite significant. CTM flow is an extracellular matrix implant that supplements and replaces damaged tissues. Small unpublished case series in total knee arthroplasty, ENT procedures, and rotator cuff repair have shown beneficial results from CTM. We hope to show similar results in this assessment of CTM in the Post-operative CMC arthroplasty patient population.

The primary outcome measure will be narcotic use postoperatively in the first 3 weeks after surgery, as measured by patient tracking. Patients will track post-op pain meds including narcotics, and OTC pain medication for the duration of their follow up period. Per standard of care, patients will be encouraged to change to Tylenol and/or ibuprofen pain medicine as soon as they are able.

Secondary outcomes will be quickDASH and VAS pain.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age 18 or older
2. Patients presenting for basilar thumb reconstruction surgery (any surgical technique)
3. Patients who can consent to be a part of this study
4. Patients who are able to return to the Indiana Hand to Shoulder Center or satellite location for follow up time points

Exclusion Criteria:

1. Additional procedures at the same time
2. Patients with previous basilar thumb reconstruction on the operative side (revision surgery)
3. Chronic narcotic use
4. Women who are pregnancy or breastfeeding
5. Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Narcotic Use | 6 Weeks
  number of narcotic medications taken in recover

SECONDARY OUTCOMES:
VAS Pain | 6 Months
  PROM
quickDASH | 6 Months
  PROM

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana Hand to Shoulder Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No